CLINICAL TRIAL: NCT05560555
Title: Tafamidis 61mg, Outcomes in ATTR Amyloidosis With Neurologic and Multisystemic Involvement - TRAMA
Brief Title: Retrospective Study Collecting Neurological Follow-up of Hereditary Transthyretin Amyloidosis (ATTRv) Patients Included in B3461028 and B3461045.
Acronym: TRAMA
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B3461104; TRAMA (Other: Alias Study Number)
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Results first posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2023-11

CONDITIONS: Hereditary Transthyretin Amyloidosis (ATTRv); Polyneuropathy
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related; Polyneuropathies | interventions — tafamidis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective cohort ATTRv and ATTRwt patients enrolled in B3461028 and B3461045 studies in Spain
  Interventions: Drug: Tafamidis

INTERVENTIONS:
Drug: Tafamidis — 61 milligrams (mg) as received in studies B3461028 and B3461045

SUMMARY:
A study of patients with hereditary transthyretin amyloidosis (ATTRv) and wild-type transthyretin amyloidosis (ATTRwt) that have been enrolled in B3461028 and B3461045 studies in Spain - exposed to tafamidis 61mg for ≥12 months with polyneuropathy (PN) have kept going to their multisystemic follow-ups (neuro/ophthalmo/gastrointestinal) ≥12 months.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with tafamidis 61 mg ≥ 12 months
* Neurological follow up ≥ 12 months
* Diagnosis of transthyretin amyloidosis with polyneuropathy (ATTR-PN) based on one of the following:
* Amplitude reduction in, at least, 2 nerves under normal value, excluding median nerve OR 50% amplitude reduction in, at least, 2 nerves on the basal value of the patient, excluding median nerve OR 2 abnormal tests detecting thin fibers alterations (through Sudo scan, RR Interval analysis, etc..)

Exclusion Criteria:

* Treatment with tafamidis 61 mg < 12 months
* Neurological follow up < 12 months
* Other diagnosis for polyneuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population: retrospective cohort of patients with hereditary transthyretin amyloidosis (ATTRv) and wild-type transthyretin amyloidosis (ATTRwt) that have been enrolled in B3461028 and B3461045 studies in Spain - exposed to tafamidis 61mg for ≥12 months with polyneuropathy have kept going to their multisystemic follow-ups (neuro/ophthalmo/gastrointestinal) ≥12 months
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2022-10-24 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (3):
- Spain (3):
  - Hospital Universitari de Bellvitge, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Son Llatzer, Palma de Mallorca

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B3461104

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with hereditary transthyretin amyloidosis (ATTRv) and wild-type transthyretin amyloidosis (ATTRwt) from studies B3461028 (NCT01994889) and B3461045 (NCT02791230) in Spain, with cardiac and neurologic exposed to Tafamidis free acid 61 milligrams (mg) for at least 12 months, and who were in neurological follow-up for no less than 12 months were observed in this retrospective study.
Pre-assignment Details: Data was collected from medical records and analyzed over 22 days of this study.
Groups:
- ATTRv: Participants diagnosed with ATTRv in studies B3461028 (NCT01994889) and B3461045 (NCT02791230) in Spain who presented with multisystem involvement (cardiac and neurological) and received tafamidis free acid 61 mg for at least 12 months were included.
- ATTRwt: Participants diagnosed with ATTRwt in studies B3461028 (NCT01994889) and B3461045 (NCT02791230) in Spain who presented with multisystem involvement (cardiac and neurological) and received tafamidis free acid 61 mg for at least 12 months were included.
Period: Overall Study
Arm/Group | ATTRv | ATTRwt
Started | 2 | 3
Completed | 2 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Groups:
- Total: Total of all reporting groups
Arm/Group | ATTRv | ATTRwt | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Continuous [Median (Full Range); unit: Years] — Age at enrollment was reported.
  Years | 71.5 [65.0 to 78.0] | 78.0 [77.0 to 79.0] | 75.4 [65.0 to 79.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 3 | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Number of participants according to Genotype [Count of Participants; unit: Participants] — Number of participants according to genotype (Mutation / Wildtype)
  Participants
    Mutation | 2 | 0 | 2
    Wild Type | 0 | 3 | 3
Age at onset of disease [Median (Full Range); unit: Years] | 67.0 [61.0 to 73.0] | 75.3 [73.0 to 77.0] | 72.0 [61.0 to 77.0]
Age at diagnosis [Median (Full Range); unit: Years] | 68.0 [61.0 to 75.0] | 77.0 [75.0 to 79.0] | 73.4 [61.0 to 79.0]
First disease-related sign or symptom [Count of Participants; unit: Participants] — Number of participants according to first disease related signs and symptoms were reported.
  Participants
    Gastrointestinal disorders | 0 | 0 | 0
    Urological disorders | 0 | 0 | 0
    Ophthalmological disorders | 0 | 0 | 0
    CNS disorders | 0 | 0 | 0
    Autonomic neuropathy changes | 1 | 2 | 3
    Peripheral neuropathy | 0 | 0 | 0
    Heart disorders | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change in Neuropathy Impairment Score (NIS) at Month 12 for ATTRv
Description: NIS (Neuropathy Impairment Score) is a clinically important, sensitive measure of individual neurological function, assessing sensory function, reflexes, and muscle weakness. NIS score ranged from 0 to 244, with higher score indicating greater disability or impairment. The rate of change was calculated from last follow-up.
Time Frame: Baseline and Month 12 (data collected and analyzed over 22 days)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Median (Full Range); unit: Change in score*months
Arm/Group | ATTRv
Number analyzed (Participants) | 2
Change in score*months | 1.6 [0.0 to 3.1]

2. Secondary Outcome: Change in NIS for ATTRv
Description: as for outcome 1
Time Frame: Baseline, Month 6, 18, 24 and 36 after the start of treatment (data collected and analyzed over 22 days)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Median (Full Range); unit: Change in score*months
Arm/Group | ATTRv
Number analyzed (Participants) | 2
Change in score*months
  Month 6 | 0.8 [0.0 to 1.6]
  Month 18 | 2.4 [0.0 to 4.7]
  Month 24 | 3.1 [0.0 to 6.3]
  Month 36 | 4.7 [0.0 to 9.4]

3. Secondary Outcome: Change in Neuropathy Impairment Score - Lower Limbs (NIS-LL) for ATTRv
Description: NIS-LL (Neuropathy Impairment Score Lower Limbs) is a clinically important, sensitive measure of neurological function in individuals, assessing sensory function, reflexes, and muscle weakness of the lower limbo. NÍS-LL assessed muscle weakness, reflexes, sensation. Each item is scored separately for left and right limbs. Components of muscle weakness:0(normal) to4(paralysis), higher score=more weakness; reflexes, sensation:0=normal, 1=decreased, or 2=absent. Total NIS-LL score range 0-88, higher score=more impairment. The rate of change was calculated from last follow-up.
Time Frame: Baseline, Month 6, 12, 18, 24 and 36 after the start of treatment (data collected and analyzed over 22 days)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Median (Full Range); unit: Change in score*months
Arm/Group | ATTRv
Number analyzed (Participants) | 1
Change in score*months
  Month 6 | 1.6 [1.6 to 1.6]
  Month 12 | 3.1 [3.1 to 3.1]
  Month 18 | 4.7 [4.7 to 4.7]
  Month 24 | 6.3 [6.3 to 6.3]
  Month 36 | 9.4 [9.4 to 9.4]

4. Secondary Outcome: Change in Norfolk Quality of Life- Diabetic Neuropathy (Norfolk QOL-DN) for ATTRv
Description: Norfolk Quality of Life Questionnaire for Diabetic Neuropathy is a standardized and validated instrument that assesses the effect of polyneuropathy on the functionality and quality of life of the individual. Norfolk QOL-DN: 35-item participant-rated questionnaire is used to assess impact of diabetic neuropathy on the quality of life of participants with diabetic neuropathy; Item 1 to 7: related to symptoms and presence of symptom was assessed as 1 and absence was assessed as 0. Item 8-35: related to activities of daily living and scored on a 5-point Likert scale, where 0= no problem and 4= severe problem (except item 32, where -2= much better, 0=about the same, 2=much worse). TQOL= sum of all the items, total possible score range= -4 to 138, where higher score=worse quality of life.
Time Frame: Baseline, Month 6, 12, 18, 24 and 36 after the start of treatment (data collected and analyzed over 22 days)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | ATTRv
Number analyzed (Participants) | 2
Units on a scale | NA [NA to NA] — Data could not be calculated due to absence of data in the records at baseline.

5. Secondary Outcome: Change in COMPASS-31 for ATTRv
Description: COMPASS-31 (Composite Autonomic Symptom Score 31) is a questionnaire designed to assess the severity and functional ability in participants with autonomic dysfunction. COMPASS-31 total score ranged from 0 to 100; where 0=Lesser severity of dysautonomia and 100=Greater severity of dysautonomia.
Time Frame: Baseline, Month 6, 12, 18, 24 and 36 after the start of treatment (data collected and analyzed over 22 days)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | ATTRv
Number analyzed (Participants) | 2
Units on a scale | NA [NA to NA] — Data could not be calculated due to absence of data in the records at baseline.

6. Secondary Outcome: Change in Familial Amyloid Polyneuropathy Specific Rasch-Built Overall Disability Scale (FAP-RODs) for ATTRv
Description: FAP-RODS is a questionnaire that assessed the effect of neuropathy on daily activities. FAP-RODS total score ranged from 0 to 68; where, 0=Lower ability to perform daily activities and 68=Greater ability to perform daily activities.
Time Frame: Baseline, Month 6, 12, 18, 24 and 36 after the start of treatment (data collected and analyzed over 22 days)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Median (Full Range); unit: Units on a scale
Arm/Group | ATTRv
Number analyzed (Participants) | 2
Units on a scale | NA [NA to NA] — Data could not be calculated due to absence of data in the records at baseline.

7. Secondary Outcome: Number of Participants According to Familiar Amyloidotic Polyneuropathy Stage (FAP) for ATTRv
Description: FAP is a stage system based on symptom severity and disease progression. FAP stages included: Asymptomatic; Free ambulation (walking without support): stage 1; Supportive ambulation (walking with support): stage 2; Wheelchair-bound or bedridden: stage 3.
Time Frame: Month 18, 24 and 30 months after the start of treatment (data collected and analyzed over 22 days)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study. Here, 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | ATTRv
Number analyzed (Participants) | 2
Participants
  Asymptomatic (Month 18): number analyzed (Participants) | 0
  Walking without support (Month 18): number analyzed (Participants) | 0
  Walking with support (Month 18): number analyzed (Participants) | 0
  Wheelchair or bedridden (Month 18): number analyzed (Participants) | 0
  Asymptomatic (Month 24): number analyzed (Participants) | 1
  Asymptomatic (Month 24) | 0
  Walking without support (Month 24): number analyzed (Participants) | 1
  Walking without support (Month 24) | 1
  Walking with support (Month 24): number analyzed (Participants) | 1
  Walking with support (Month 24) | 0
  Wheelchair or bedridden (Month 24): number analyzed (Participants) | 1
  Wheelchair or bedridden (Month 24) | 0
  Asymptomatic (Month 30) | 1
  Walking without support (Month 30) | 1
  Walking with support (Month 30) | 0
  Wheelchair or bedridden (Month 30) | 0

8. Secondary Outcome: Percentage of Participants Who do Not Have Stage Progression in the PND Score for ATTRv
Description: PND is a staging system that assess the degree of neuropathic dysfunction and its impact on ambulation. PND stages included: Asymptomatic; Stage I: Sensory disturbances, normal gait; Stage II: Sensory disturbances, altered gait not requiring support; IIIA: Gait requiring one support; IIIB: Gait requiring two supports; IV: Wheelchair or bedside. Participants who did not change to higher stages compared to the start of treatment was reported as Unchanged and those who progressed to higher stages were reported under Staging up.
Time Frame: From Baseline to Month 30 (data collected and analyzed over 22 days)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Number; unit: Percentage of participants
Arm/Group | ATTRv
Number analyzed (Participants) | 2
Percentage of participants
  Unchanged | 100.0
  Staging up | 0.0

9. Secondary Outcome: Percentage of Responders to Treatment for ATTRv
Description: Percentage of responders to treatment at Month 12 was defined as participants who achieved the change from baseline of less than 4 points in the NIS and participants who achieved the change from baseline of less than 2 points in the NIS-LL were reported in this outcome measure.
Time Frame: Month 12 (data collected and analyzed over 22 days)
Population: as for outcome 7
Measure: Number; unit: Percentage of responders
Arm/Group | ATTRv
Number analyzed (Participants) | 2
Percentage of responders
  NIS | 100.0
  NIS-LL: number analyzed (Participants) | 1
  NIS-LL | 0.0

10. Secondary Outcome: Number of Participants With R-R Interval Variability for ATTRv
Description: Number of participants with R-R interval variability (altered/unaltered) was reported in this outcome measure.
Time Frame: Month 18, 24 and 30 (data collected and analyzed over 22 days)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure. 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | ATTRv
Number analyzed (Participants) | 1
Participants
  Unaltered (Month 18): number analyzed (Participants) | 0
  Altered (Month 18): number analyzed (Participants) | 0
  Unaltered (Month 24): number analyzed (Participants) | 0
  Altered (Month 24): number analyzed (Participants) | 0
  Unaltered (Month 30) | 0
  Altered (Month 30) | 1

11. Secondary Outcome: Modified Body Mass Index (mBMI) for ATTRv
Description: BMI was calculated by weight divided by height squared and measured as kilogram per square meter (kg/m^2). mBMI was calculated by multiplying BMI by serum albumin levels [gram/liter (g/L)].
Time Frame: Month 18, 24 and 30 after start of treatment (data collected and analysed over 22 days)
Population: as for outcome 10
Measure: Median (Full Range); unit: Kilogram per meter square*gram/Liter
Arm/Group | ATTRv
Number analyzed (Participants) | 1
Kilogram per meter square*gram/Liter
  Month 18: number analyzed (Participants) | 0
  Month 24 | 27.7 [27.7 to 27.7]
  Month 30 | 24.3 [24.3 to 24.3]

12. Secondary Outcome: Ulnar/Sural Sensory Nerve Action Potential Amplitude (SNAP) for ATTRv
Description: Sural sensory nerve action potential amplitude (in microvolts) was measured using electromyography of the left lower limb.
Time Frame: Month 24 and 30 after the start of treatment (data collected and analyzed over 22 days)
Population: as for outcome 7
Measure: Median (Full Range); unit: Micro volts (μV)
Arm/Group | ATTRv
Number analyzed (Participants) | 2
Micro volts (μV)
  Month 24: number analyzed (Participants) | 0
  Month 30 | 2.9 [1.1 to 4.6]

13. Secondary Outcome: Ulnar/Peroneal Compound Muscle Action Potential Amplitude (CMAP) for ATTRv
Description: Peroneal motor nerve compound muscle action potential amplitude was measured using electromyography of the left lower limb.
Time Frame: Month 24 and 30 after the start of treatment (data collected and analyzed over 22 days)
Population: as for outcome 7
Measure: Median (Full Range); unit: Milli Volts (mV)
Arm/Group | ATTRv
Number analyzed (Participants) | 2
Milli Volts (mV)
  Month 24: number analyzed (Participants) | 0
  Month 30 | 1.3 [1.1 to 1.5]

14. Secondary Outcome: Change in NIS for ATTRwt
Description: NIS (Neuropathy Impairment Score) was a clinically important, sensitive measure of individual neurological function, assessing sensory function, reflexes, and muscle weakness. NIS score ranged from 0 to 244, with higher score indicating greater disability or impairment. The rate of change was calculated from last follow-up.
Time Frame: Baseline, Month 6, 12, 18, 24 and 36 after the start of treatment (data collected and analyzed over 22 days)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Median (Full Range); unit: Change in score*months
Arm/Group | ATTRwt
Number analyzed (Participants) | 3
Change in score*months
  Month 6 | 0.4 [0.0 to 0.8]
  Month 12 | 0.8 [0.0 to 1.5]
  Month 18 | 1.1 [0.0 to 2.3]
  Month 24 | 1.5 [0.0 to 3.0]
  Month 36 | 2.3 [0.0 to 4.5]

15. Secondary Outcome: Change in NIS-LL for ATTRwt
Description: NIS-LL (Neuropathy Impairment Score Lower Limbs) was clinically important, sensitive measure of neurological function in individuals, assessing sensory function, reflexes, and muscle weakness of the lower limbo. NÍS-LL assessed muscle weakness, reflexes, sensation. Each item scored separately for left and right limbs. Components of muscle weakness:0(normal) to4(paralysis), higher score=more weakness; reflexes, sensation:0=normal, 1=decreased, or 2=absent. Total NIS-LL score range 0-88, higher score=more impairment. The rate of change was calculated from last follow-up.
Time Frame: Baseline, Month 6, 12, 18, 24 and 36 after the start of treatment (data collected and analyzed over 22 days)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Median (Full Range); unit: Change in score*months
Arm/Group | ATTRwt
Number analyzed (Participants) | 2
Change in score*months
  Month 6 | 0.2 [0.0 to 0.4]
  Month 12 | 0.4 [0.0 to 0.8]
  Month 18 | 0.6 [0.0 to 1.2]
  Month 24 | 0.8 [0.0 to 1.6]
  Month 36 | 1.2 [0.0 to 2.3]

16. Secondary Outcome: Change in Norfolk QOL-DN for ATTRwt
Description: Norfolk Quality of Life Questionnaire for Diabetic Neuropathy was a standardized and validated instrument that assesses the effect of polyneuropathy on the functionality and quality of life of the individual. Norfolk QOL-DN: 35-item participant-rated questionnaire used to assess impact of diabetic neuropathy on the quality of life of participants with diabetic neuropathy; Item 1 to 7: related to symptoms and presence of symptom was assessed as 1 and absence was assessed as 0. Item 8-35: related to activities of daily living and scored on a 5-point Likert scale, where 0= no problem and 4= severe problem (except item 32, where -2= much better, 0=about the same, 2=much worse). TQOL= sum of all the items, total possible score range= -4 to 138, where higher score=worse quality of life.
Time Frame: Baseline, Month 6, 12, 18, 24 and 36 after the start of treatment (data collected and analyzed over 22 days)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study. Data was not collected for this outcome measure as data was not available in the medical records.
Arm/Group | ATTRwt
Number analyzed (Participants) | 0

17. Secondary Outcome: Change in COMPASS-31 for ATTRwt
Description: COMPASS-31 (Composite Autonomic Symptom Score 31) was a questionnaire designed to assess the severity and functional ability in participants with autonomic dysfunction. COMPASS-31 total score ranged from 0 to 100; where 0=Lesser severity of dysautonomia and 100=Greater severity of dysautonomia.
Time Frame: Baseline, Month 6, 12, 18, 24 and 36 after treatment initiation
Population: as for outcome 16
Arm/Group | ATTRwt
Number analyzed (Participants) | 0

18. Secondary Outcome: Change in FAP-RODs for ATTRwt
Description: as for outcome 6
Time Frame: Baseline, Month 6, 12, 18, 24 and 36 after the start of treatment (data collected and analyzed over 22 days)
Population: as for outcome 16
Arm/Group | ATTRwt
Number analyzed (Participants) | 0

19. Secondary Outcome: Number of Participants According to FAP Stage for ATTRwt
Description: FAP stage is a staging system based on symptom severity and disease progression. FAP stages included: Asymptomatic; Free ambulation (Walking without support): stage 1; Supportive ambulation (Walking with support): stage 2; Wheelchair-bound or bedridden: stage 3.
Time Frame: Month 18, 24 and 30 months after the start of treatment (data collected and analyzed over 22 days)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | ATTRwt
Number analyzed (Participants) | 2
Participants
  Asymptomatic (Month 18): number analyzed (Participants) | 1
  Asymptomatic (Month 18) | 0
  Walking without support (Month 18): number analyzed (Participants) | 1
  Walking without support (Month 18) | 1
  Walking with support (Month 18): number analyzed (Participants) | 1
  Walking with support (Month 18) | 0
  Wheelchair or bedridden (Month 18): number analyzed (Participants) | 1
  Wheelchair or bedridden (Month 18) | 0
  Asymptomatic (Month 24) | 0
  Walking without support (Month 24) | 2
  Walking with support (Month 24) | 0
  Wheelchair or bedridden (Month 24) | 0
  Asymptomatic (Month 30) | 0
  Walking without support (Month 30) | 2
  Walking with support (Month 30) | 0
  Wheelchair or bedridden (Month 30) | 0

20. Secondary Outcome: Percentage of Participants Who do Not Have Stage Progression in the PND Score for ATTRwt
Description: PND was a simple staging system according to the degree of neuropathic dysfunction and its impact on ambulation. PND stages included: Asymptomatic: I Sensory disturbances, normal gait: II Sensory disturbances, altered gait not requiring support: IIIA Gait requiring one support: IIIB Gait requiring two supports: IV Wheelchair or bedside). Participants who did not change to higher stages compared to the start of treatment was reported as Unchanged and those who progressed to higher stages were reported under Staging up.
Time Frame: From Baseline to Month 30 (data collected and analysed over 22 days)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Number; unit: Percentage of participants
Arm/Group | ATTRwt
Number analyzed (Participants) | 3
Percentage of participants
  Unchanged | 66.7
  Staging up | 33.3

21. Secondary Outcome: Percentage of Responders to Treatment for ATTRwt
Description: Percentage of responders to treatment was defined as participants who achieved the change from baseline of less than 4 points in the NIS and participants who achieved the change from baseline of less than 2 points in the NIS-LL were reported in this outcome measure.
Time Frame: Month 12 (data collected and analyzed over 22 days)
Population: as for outcome 7
Measure: Number; unit: Percentage of responders
Arm/Group | ATTRwt
Number analyzed (Participants) | 3
Percentage of responders
  NIS | 100.0
  NIS-LL: number analyzed (Participants) | 2
  NIS-LL | 100.0

22. Secondary Outcome: Number of Participants With R-R Interval Variability for ATTRwt
Description: Number of participants with R-R interval variability (altered/unaltered) was reported in this outcome measure.
Time Frame: Month 18, 24 and 30 (data collected and analyzed over 22 days)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | ATTRwt
Number analyzed (Participants) | 1
Participants
  Unaltered (Month 18): number analyzed (Participants) | 0
  Altered (Month 18): number analyzed (Participants) | 0
  Unaltered (Month 24) | 0
  Altered (Month 24) | 1
  Unaltered (Month 30) | 0
  Altered (Month 30) | 1

23. Secondary Outcome: mBMI for ATTRwt
Description: BMI was calculated by weight divided by height squared and measured as kilogram per square meter (kg/m^2).
Time Frame: Month 18, 24 and 30 after start of treatment (data collected and analysed over 22 days)
Population: as for outcome 10
Measure: Median (Full Range); unit: Kilogram per meter square*gram/Liter
Arm/Group | ATTRwt
Number analyzed (Participants) | 2
Kilogram per meter square*gram/Liter
  Month 18: number analyzed (Participants) | 1
  Month 18 | 29.7 [29.7 to 29.7]
  Month 24 | 24.0 [22.1 to 26.0]
  Month 30 | 25.7 [22.1 to 29.4]

24. Secondary Outcome: Ulnar/Sural SNAP Score for ATTRwt
Description: as for outcome 12
Time Frame: Month 24 and 30 after the start of treatment (data collected and analyzed over 22 days)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study. Here, 'Overall Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Median (Full Range); unit: Micro volts (μV)
Arm/Group | ATTRwt
Number analyzed (Participants) | 1
Micro volts (μV)
  Month 24 | 17.0 [17.0 to 17.0]
  Month 30 | 11.9 [11.9 to 11.9]

25. Secondary Outcome: Ulnar/Peroneal CMAP Score for ATTRwt
Description: Peroneal motor nerve compound muscle action potential amplitude (in millivolts) was measured using electromyography of the left lower limb.
Time Frame: Month 24 and 30 after the start of treatment (data collected and analyzed over 22 days)
Population: as for outcome 24
Measure: Median (Full Range); unit: Milli Volts (mV)
Arm/Group | ATTRwt
Number analyzed (Participants) | 1
Milli Volts (mV)
  Month 24 | 5.9 [5.9 to 5.9]
  Month 30 | 2.7 [2.7 to 2.7]

26. Secondary Outcome: Number of Participants With Carpal Tunnel Syndrome
Description: Number of participants with carpal tunnel syndrome were reported in this outcome measure.
Time Frame: At baseline (data collected and analyzed over 22 days)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | ATTRv | ATTRwt
Number analyzed (Participants) | 2 | 3
Participants | 2 | 2

27. Secondary Outcome: Number of Participants With Lumbar Stenosis
Description: Number of participants with lumbar stenosis were reported in this outcome measure.
Time Frame: At baseline (data collected and analyzed over 22 days)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | ATTRv | ATTRwt
Number analyzed (Participants) | 2 | 3
Participants | 0 | 1

28. Secondary Outcome: Number of Participants With Gastrointestinal Disturbances
Description: Number of participants with gastrointestinal disturbances were reported in this outcome measure.
Time Frame: Month 18, 24 and 30 after the start of treatment (data collected and analyzed over 22 days)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | ATTRv | ATTRwt
Number analyzed (Participants) | 2 | 3
Participants
  Month 18: number analyzed (Participants) | 0 | 1
  Month 18 |  | 1
  Month 24: number analyzed (Participants) | 1 | 2
  Month 24 | 0 | 1
  Month 30: number analyzed (Participants) | 2 | 2
  Month 30 | 0 | 2

29. Secondary Outcome: Number of Participants With Unintentional Weight Loss
Description: Number of participants with unintentional weight loss were reported in this outcome measure.
Time Frame: Month 18, 24 and 30 after the start of treatment (data collected and analyzed over 22 days)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study. Here, 'Overall Number Analyzed' signifies participants evaluable for this outcome measure and 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | ATTRv | ATTRwt
Number analyzed (Participants) | 0 | 2
Participants
  Month 18: number analyzed (Participants) | 0 | 1
  Month 18 |  | 0
  Month 24: number analyzed (Participants) | 0 | 1
  Month 24 |  | 0
  Month 30 |  | 0

30. Secondary Outcome: Number of Participants With Urological Disturbances
Description: Number of participants with urological disturbances were reported in this outcome measure.
Time Frame: Month 18, 24 and 30 after the start of treatment (data collected and analyzed over 22 days)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study. All participants in the 'Overall Number of Participants Analyzed' contributed data to the table but may not have evaluable data for every row. Here, 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | ATTRv | ATTRwt
Number analyzed (Participants) | 2 | 3
Participants
  Month 18: number analyzed (Participants) | 0 | 1
  Month 18 | 0 | 0
  Month 24: number analyzed (Participants) | 1 | 2
  Month 24 | 0 | 0
  Month 30: number analyzed (Participants) | 2 | 2
  Month 30 | 0 | 1

31. Secondary Outcome: Number of Participants With Ophthalmological Disturbances
Description: Number of participants with ophthalmological disturbances were reported in this outcome measure.
Time Frame: Month 18, 24 and 30 after the start of treatment (data collected and analyzed over 22 days)
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | ATTRv | ATTRwt
Number analyzed (Participants) | 2 | 3
Participants
  Month 18: number analyzed (Participants) | 0 | 1
  Month 18 | 0 | 0
  Month 24: number analyzed (Participants) | 1 | 2
  Month 24 | 0 | 0
  Month 30: number analyzed (Participants) | 2 | 2
  Month 30 | 0 | 0

32. Secondary Outcome: Number of Participants With Central Nervous System (CNS) Disturbances
Description: Number of participants with CNS disturbances were reported in this outcome measure.
Time Frame: Month 18, 24 and 30 after the start of treatment (data collected and analyzed over 22 days)
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | ATTRv | ATTRwt
Number analyzed (Participants) | 2 | 3
Participants
  Month 18: number analyzed (Participants) | 0 | 1
  Month 18 | 0 | 0
  Month 24: number analyzed (Participants) | 1 | 2
  Month 24 | 0 | 0
  Month 30: number analyzed (Participants) | 2 | 2
  Month 30 | 0 | 0

33. Secondary Outcome: Number of Participants With Symptoms of Autonomic Neuropathy
Description: Number of participants with symptoms of autonomic neuropathy including impaired sweating, sexual dysfunction, orthostatic hypotension were reported in this outcome measure.
Time Frame: Month 18, 24 and 30 after the start of treatment (data collected and analyzed over 22 days)
Population: as for outcome 30
Measure: Count of Participants; unit: Participants
Arm/Group | ATTRv | ATTRwt
Number analyzed (Participants) | 2 | 2
Participants
  Month 18: number analyzed (Participants) | 0 | 1
  Month 18 | 0 | 1
  Month 24: number analyzed (Participants) | 1 | 2
  Month 24 | 0 | 2
  Month 30 | 1 | 2

34. Secondary Outcome: Number of Participants With Symptoms of Peripheral Neuropathy
Description: Number of participants with symptoms of peripheral neuropathy (allodynia and paresthesia) were reported in this outcome measure.
Time Frame: At baseline (data collected and analyzed over 22 days)
Population: Analysis population included all eligible participants whose data was retrieved and analyzed in this study.
Measure: Count of Participants; unit: Participants
Arm/Group | ATTRv | ATTRwt
Number analyzed (Participants) | 2 | 3
Participants | 1 | 0

ADVERSE EVENTS:
Time Frame: From start of treatment until Month 36 (data collected and analyzed over 22 days)
Arm/Group | ATTRv | ATTRwt
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 0/2 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-02-17): https://cdn.clinicaltrials.gov/large-docs/55/NCT05560555/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/55/NCT05560555/SAP_001.pdf